CLINICAL TRIAL: NCT06769464
Title: Electrophysiological Representations of Odor in the Human Brain Study 1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Christina Zelano, Associate Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 60067814-1
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Odor Intensity Ratings
MeSH Terms: interventions — Odorants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigating representations of odor intensity in human piriform cortex. (Experimental): Odors will be presented at different concentrations.
  Interventions: Behavioral: odor

INTERVENTIONS:
Behavioral: odor — present odor

SUMMARY:
Investigating representations of odor intensity in human piriform cortex. To identify a neural representation of perceived odor intensity, it is necessary to dissociate stimulus concentration from perceived intensity. Experiments for this aim will measure human perceptual responses while manipulating intensity independently from concentration using two complementary approaches. In Experiment 1A, we will match perceived intensities across odors of different concentrations, allowing us to identify a neural representation of intensity that is independent of stimulus identity and concentration. In Experiment 1B, we will create conditions of different perceived intensity over constant odor stimuli using adaptation. Approaching the same question from different angles will strengthen the robustness of our findings. Preliminary data suggest that temporal features of the piriform neural response may represent odor intensity.

DETAILED DESCRIPTION:
Olfactory perception relies on the brain's ability to extract and represent different features of an odor stimulus. For example, intensity and identity are fundamental features of the olfactory percept that must be encoded separately for accurate perception; the same odor can be encountered at different strengths. Understanding neural representations of olfactory perceptual features is fundamental to understanding the olfactory system, however the neural correlates of odor intensity and identity are poorly understood in the human brain.

The field of olfaction typically uses chemistry as a proxy for perception and focuses on manipulating physical properties of a stimulus to look for neural correlates. For example, chemical concentration and molecular identity are typically used as proxies for odor intensity and identity. However, the world that animals perceive is not a complete representation of physical reality; it is a product of the particular sensory systems that each species has acquired in the course of evolution. To understand how the brain forms representations of perceptual features of odors, we must identify relationships between features of neural responses and perceptual ratings. While novel behavioral paradigms in rodents can provide good estimates of perceptual ratings of different features of odors (intensity, identity), humans can directly provide perceptual ratings of different features of an odor. Therefore, human work is necessary to fully understand olfactory perception.

The missing link between neural signatures and perceptual properties of odor is a critical gap in our understanding of odor coding. Here, we will combine human intracranial recordings-including direct neural recordings from human olfactory cortex-with simultaneous delivery of precisely controlled odors of varying intensity/identity and trial-by-trial collection of psychophysical ratings to understand how odors are represented in the human brain.

Accurate olfactory psychophysical ratings are a critical part of our proposal. Therefore, we will work with leading experts in human psychophysics at Monel Chemical Senses Center, Dr. Pamela Dalton and Dr. Joel Mainland. As Co-Investigators on this grant, their expertise in human psychophysics will combine with my lab's expertise in human olfactory electrophysiology to provide the field with an understanding of the mappings between olfactory perception and neural codes in the human brain.

Aim 1: Investigating representations of odor intensity in human piriform cortex. To identify a neural representation of perceived odor intensity, it is necessary to dissociate stimulus concentration from perceived intensity. Experiments for this aim will measure human perceptual responses while manipulating intensity independently from concentration using two complementary approaches. In Experiment 1A, we will match perceived intensities across odors of different concentrations, allowing us to identify a neural representation of intensity that is independent of stimulus identity and concentration. In Experiment 1B, we will create conditions of different perceived intensity over constant odor stimuli using adaptation. Approaching the same question from different angles will strengthen the robustness of our findings. Preliminary data suggest that temporal features of the piriform neural response may represent odor intensity.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12 to 65, english speaker, patients undergoing brain surgery for treatment of medically intractable epilepsy

Exclusion Criteria:

* screening for history of smell or taste problems

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Perceived odor intensity | 15 minutes
  Odors of different concentrations will be presented, and we will obtain behavioral ratings on a GLMS scale of intensity presented on a laptop computer, converted into Matlab for analysis

CONTACTS AND LOCATIONS:
Overall Officials: christina zelano, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States